CLINICAL TRIAL: NCT04077515
Title: Safety and Efficacy of Low-dose Sirolimus to Kaposiform Hemangioendothelioma:A Prospective, Randomized Open Trial
Brief Title: Safety and Efficacy of Low-dose Sirolimus to Kaposiform Hemangioendothelioma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-161
Record Dates: First submitted 2019-06-25; First posted 2019-09-04 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Hemangioma; Kaposiform Hemangioendothelioma
Keywords: Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome; Sirolimus; Rapamycin
MeSH Terms: conditions — Hemangioma; Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high blood concentration group (Active Comparator): The blood concentration is maintained at 10-15ng/ml (not including 10ng/ml).
  Interventions: Drug: Sirolimus(0.8mg/m2)
- low blood concentration group (Experimental): The blood concentration is maintained at 7-10ng/ml (including 10ng/ml).
  Interventions: Drug: Sirolimus(0.7mg/m2)

INTERVENTIONS:
Drug: Sirolimus(0.8mg/m2) — The initial use of sirolimus is 0.8mg/m2 administered twice daily.After two weeks of taking the drug, blood concentrations are measured and adjusted appropriately to maintain the targeted blood concentration.
  Other Names: Rapamycin
  Arms: high blood concentration group
Drug: Sirolimus(0.7mg/m2) — The initial use of sirolimus is 0.7mg/m2 administered twice daily.After two weeks of taking the drug, blood concentrations are measured and adjusted appropriately to maintain the targeted blood concentration.
  Other Names: Rapamycin
  Arms: low blood concentration group

SUMMARY:
to evaluate the safety and efficacy of Low-dose sirolimus in Kaposiform Hemangioendothelioma in Chinese children by a prospective, randomized open trial.

DETAILED DESCRIPTION:
The clinically commonly used dose of sirolimus for Kaposiform Hemangioendothelioma is 0.8 mg/m2 administered twice daily, and the blood concentration can be maintained at 10-15 ng/ml according to the pharmacokinetic formula.Related research reports that maintaining low blood concentration of sirolimus is effective in the treatment of certain vascular malformations and hemangioma, and complications are less. In the clinical practice, we found that the blood concentration was maintained at 7-10 ng/ml, and the patients still achieved good results and the chance of infections decreased. Therefore, this clinical trial was designed.In this trial, two different dosing regimens with corresponding blood concentration were designed to compare the safety and efficacy.In the high concentration group, the sirolimus dosage was adjusted monthly to achieve trough levels between 10 and 15 ng/mL(excluding 10 ng/ml), and it is still used at 0.8 mg/m2 administered twice daily.The low concentration group is 7-10 ng/ml (including 10 ng/ml), and the initial use of sirolimus is 0.7mg/m2 administered twice daily.The dose was adjusted according to the formula after two weeks.The follow-up and evaluation were performed according to a strictly established follow-up schedule after taking the drug.

ELIGIBILITY:
Inclusion Criteria:

* Kaposiform Hemangioendotheliomas with or without Kasabach-Merritt Phenomenon.
* 0 - 12 years of age at the time of study entry.
* Male or female.
* Consent of parents (or the person having parental authority in families): Signed and dated written informed consent.

Exclusion Criteria:

* with hematological diseases.
* with other solid tumors.
* with hypertension, diabetes, adrenal insufficiency, neurological diseases, liver and kidney dysfunction, and cardiopulmonary insufficiency.
* with tuberculosis,cytomegalovirus and Epstein-Barr virus infection before the treatment.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
response to treatment | 1 year after taking the drug
  it is a variable outcome, including complete responses, partial response and no response.
  The definitions are :
  Complete Response：
  1. platelets counts is greater than 100×10^9/L.
  2. significant volume reduction is greater than 80%.
  3. Fibrinogen levels at 2-4g/L.
  4. The surface skin of the tumor is lighter or the tumor is softer significantly.
  Partial Response:
  1. platelets counts is greater than 40×10^9/L.
  2. significant volume reduction is greater than 50%.
  3. Fibrinogen levels at less than 50% reduction from baseline.
  4. The surface skin of the tumor and palpation of the tumor have no change or less change.
  No Response:
  1. platelets counts is less than 40×10^9/L.
  2. significant volume reduction is less than 50% or the tumor is bigger.
  3. Fibrinogen levels at grater then 50% reduction from baseline.
  4. The surface skin of the tumor is darker or the tumor is harder.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year after taking the drug
  Monitoring patient's clinical biochemical indicators and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drolet BA, Trenor CC 3rd, Brandao LR, Chiu YE, Chun RH, Dasgupta R, Garzon MC, Hammill AM, Johnson CM, Tlougan B, Blei F, David M, Elluru R, Frieden IJ, Friedlander SF, Iacobas I, Jensen JN, King DM, Lee MT, Nelson S, Patel M, Pope E, Powell J, Seefeldt M, Siegel DH, Kelly M, Adams DM. Consensus-derived practice standards plan for complicated Kaposiform hemangioendothelioma. J Pediatr. 2013 Jul;163(1):285-91. doi: 10.1016/j.jpeds.2013.03.080. No abstract available. PMID 23796341
- [Background] Yoon HY, Hwang JJ, Kim DS, Song JW. Efficacy and safety of low-dose Sirolimus in Lymphangioleiomyomatosis. Orphanet J Rare Dis. 2018 Nov 14;13(1):204. doi: 10.1186/s13023-018-0946-8. PMID 30428897
- [Background] Kazmierczak D, Maliszewska A. [Disturbances of tooth and maxillary development in Down's syndrome and their treatment]. Czas Stomatol. 1986 Nov;39(11):755-9. No abstract available. Polish. PMID 2958244
- [Background] Ozgonenel B, Martin A. Low-dose sirolimus controls recurrent iron deficiency in a patient with blue rubber bleb nevus syndrome. Pediatr Blood Cancer. 2015 Nov;62(11):2054-5. doi: 10.1002/pbc.25590. Epub 2015 Jul 1. No abstract available. PMID 26132912